CLINICAL TRIAL: NCT05128747
Title: Effectiveness of Nutritional Program Intervention for Control of Lipid Profile Among Diabetic Patients
Brief Title: Effectiveness of Nutritional Program Among Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad M Galal, Principal Investigator, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Eonpifcolpadp
Record Dates: First submitted 2021-09-15; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Dyslipidemia Associated With Type II Diabetes Mellitus
MeSH Terms: interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Intervention Model Description: diabetic patients type2 with dyslipidemia
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of intervention will receive nutritional program (Active Comparator): group of type 2 diabetes on diabetic diet undergo nutritional program (low fat contents) to control the lipid profile (lowering cholesterol profile) in duration of 3 months.
  Interventions: Other: DASH diet
- group of control will not receive nutritional program (No Intervention): group of type 2 diabetes on diabetic drugs without nutritional program to compare their lipid profile with the diabetic patients on nutritional program.

INTERVENTIONS:
Other: DASH diet — it will be face to face about the role of nutritional program to control dyslipidemia
  Arms: group of intervention will receive nutritional program

SUMMARY:
Dyslipidemia is very common in type 2 diabetes mellitus affecting around 72%-85% of diabetic patients.The exact mechanism of lipoprotein abnormalities in diabetes is not very well understood. Insulin resistance, rather than hyperglycemia, has been implicated in the pathogenesis of diabetic dyslipidemia because lipoprotein changes including an increase in triglycerides (TG), increase in VLDL particles, small dense LDL particles and a decrease in HDL level have been shown in patients with impaired fasting glucose and impaired glucose tolerance and T2DM

DETAILED DESCRIPTION:
Hypertriglyceridaemia(HTG) occurs due to both increased production and decreased clearance, and it is the most common abnormality of diabetic dyslipidemia. Insulin resistance causes increased production of VLDL . In addition to increased secretion of VLDL, there is decreased clearance of VLDL due to decreased hepatic uptake and impaired activity of lipoprotein lipase.Management of dyslipidemia in patients with diabetes is an important step in the prevention of cardiovascular disease, the most common cause of death in the diabetic population. Diabetic dyslipidemia treatments can be divided into non-pharmacological and pharmacological. Non-pharmacological treatment includes ; medical nutrition therapy, weight loss, and physical activity. Diabetic patients should increase the intake of plant stanols/sterols, viscous fiber (legumes, citrus, oats), n-3 fatty acids and decrease the intake of saturated and trans-fatty acids. American Diabetes Association recommends the Mediterranean diet or DASH (Dietary Approaches to Stop Hypertension).

ELIGIBILITY:
Inclusion Criteria:

* 1-clinical diagosis of type2diabetes 2-clinical diagnosis of hyperlpidemia 3-must be helpful patient 4-age below 70year

Exclusion Criteria:

1-insulin dependant diabetes 2- pregnancy 3-heart disease 4- renal disease. 5-pregnancy

-

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of one of the most common dietary approches;DASH diet in controlling lipid profile in diabetic patients. | 3-6 months
  number of type 2 diabetic patients will undergo nutritional program to control their lipid profile to improve the insulin sensitivity and follow up the result of the diet by investigations (lipid profile) in duration 3 months .

REFERENCES:
- [Background] Jialal I, Singh G. Management of diabetic dyslipidemia: An update. World J Diabetes. 2019 May 15;10(5):280-290. doi: 10.4239/wjd.v10.i5.280. PMID 31139315
- [Background] Haffner SM, Lehto S, Ronnemaa T, Pyorala K, Laakso M. Mortality from coronary heart disease in subjects with type 2 diabetes and in nondiabetic subjects with and without prior myocardial infarction. N Engl J Med. 1998 Jul 23;339(4):229-34. doi: 10.1056/NEJM199807233390404. PMID 9673301
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Sharifirad G, Entezari MH, Kamran A, Azadbakht L. The effectiveness of nutritional education on the knowledge of diabetic patients using the health belief model. J Res Med Sci. 2009 Jan;14(1):1-6. PMID 21772854